CLINICAL TRIAL: NCT03154411
Title: A Phase 0 Open Label, Single-center Clinical Trial of ABY-029, an Anti-EGFR Fluorescence Imaging Agent Via Single Intravenous Injection to Subjects With Primary Sarcoma.
Brief Title: A Microdose Evaluation Study of ABY-029 in Primary Sarcoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Eric R. Henderson, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D16143
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Primary Soft-tissue Sarcoma
Keywords: ABY-029; Affibody; molecular fluorescence-guided surgery; Epidermal Growth Factor Receptor (EGFR)
MeSH Terms: interventions — ABY-029

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABY-029 (Experimental): ABY-029 will be administered prior to surgery and tissue will be examined ex vivo to determine binding with EGFR positive tumor tissue.
  Interventions: Drug: ABY-029

INTERVENTIONS:
Drug: ABY-029 — A minimum of 6 and a maximum of 12 adult patients with a diagnosis of primary soft-tissue sarcoma will be enrolled. Initial diagnostic biopsy specimens will be analyzed for EGFR positivity (an EGFR pathology score ≥ 1) by immunohistochemistry following routine diagnostic processing by Pathologist. Patients will be administered a single intravenous dose of ABY-029 1-3 hours before surgery.
  Other Names: ABY-029 trifluoroacetate salt; IRDye® 800CW Maleimide labeled Affibody peptide

SUMMARY:
The primary study objective is to determine if microdoses of ABY-029 (up to 6X) lead to detectable signals (defined as signal-to-noise ratio, SNR ≥10, with the Odyssey NIR scanner in sampled tissues with an EGFR pathology score ≥ 1 based on histological staining and compare SNR to tissues with an EGFR pathology score < 1).

The secondary study objective is to assess if the spatial patterns of EGFR expression correlate with the tumor targeting of ABY-029 detection by NIR scanner relative to histopathology diagnosis, and other indicators (e.g. proliferation, infiltration, etc.) as the gold standard, and to measure the molecular uptake and concentration of ABY-029 in resected specimens.

DETAILED DESCRIPTION:
The investigators plan to enroll a minimum of 6 and a maximum of 12 adult patients with a diagnosis of primary soft-tissue sarcoma in this open label, single center, clinical trial of ABY-029. The study will enroll patients with an EGFR pathology score ≥ 1.

Initial diagnostic biopsy specimens will be analyzed for EGFR positivity by immunohistochemistry following routine diagnostic processing by Pathologist. Patients will be administered a single intravenous dose of ABY-029 1-3 hours before surgery. Following tumor excision, the tumor will be transported to the Pathologist and will be inked and sectioned. Following sectioning the tumor will be imaged using near-infrared imaging systems. Quantitative measurements of fluorophore concentration will be measured for tumors with EGFR pathology score ≥ 1 and compared to those with EGFR pathology score < 1. Quantitative mapping of fluorophore concentration will be correlated with local EGFR concentration and blood vessel density. Upon specimen analysis, fluorophore measurements will be taken from normal, marginal tissues (e.g. skeletal muscle, adipose) in addition to the tumor. Average EGFR concentration and blood vessel density will be determined for each tumor through histological analysis of sections by routine sarcoma protocol and analysis guided by regional variations in ABY-029 concentration based upon near-infrared scan results.

The protocol is not a safety study since no physiological effects are expected at microdose levels of ABY-029. No diagnostic or therapeutic intent is proposed, and administration of the study drug is not intended to alter the extent of planned tumor resection during the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative histological diagnosis of primary sarcoma.
2. Tumor judged to be suitable for open surgical resection based on preoperative imaging studies.
3. Valid informed consent by subject.
4. Age ≥ 18 years old.

Exclusion Criteria:

1. Pregnant women or women who are breast feeding.
2. Patients on any experimental anti-EGFR targeted therapies, either investigational or FDA approved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Signal detection | Day of surgery, up to 1 week after surgery
  Following tumor excision, the tumor will be inked and sectioned and imaged using a near-infrared scanner and fiber-probe based system. Quantitative measurements of fluorophore concentration will be measured for tumors with EGFR pathology score ≥ 1 and compared to those with EGFR pathology score < 1.

SECONDARY OUTCOMES:
Correlation of spatial patterns of EGFR expression | within 1 week of surgery
  Quantitative mapping of fluorophore concentration will be correlated with local EGFR concentration and blood vessel density.
molecular uptake and ABY-029 concentration | within 1 week of surgery
  Fluorophore measurements will be taken from normal, marginal tissues (e.g. skeletal muscle, adipose) in addition to the tumor. Average EGFR concentration and blood vessel density will be determined for each tumor through histological analysis of sections by routine sarcoma protocol and analysis guided by regional variations in ABY-029 concentration based upon near-infrared scan results.

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Henderson, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT03154411/ICF_000.pdf